CLINICAL TRIAL: NCT04000373
Title: Pilot Study of Powered Exoskeleton Use for Gait Rehabilitation in Individuals With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Francois Bethoux, MD, Director of Rehabilitation Services at the Cleveland Clinic Mellen Center., The Cleveland Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-580
Record Dates: First submitted 2019-06-06; First posted 2019-06-27 (Actual); Results first posted 2020-04-07 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Multiple Sclerosis; Gait Disorders, Neurologic
MeSH Terms: conditions — Multiple Sclerosis; Gait Disorders, Neurologic

STUDY DESIGN:
Intervention Model Description: uncontrolled pre-post intervention study of the use of the Ekso GT™exoskeleton in gait training in the MS population
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- gait training with exoskeleton device (Other): uncontrolled pre-post intervention study of gait training using the Ekso GT™exoskeleton
  Interventions: Device: Ekso GT™ exoskeleton

INTERVENTIONS:
Device: Ekso GT™ exoskeleton — The rehabilitation treatment will consist of 3 sessions per week for 8 weeks, for a total of 24 sessions. Missed sessions will be made up if possible. Each session will be scheduled for 60 minutes, and will consist of stretching, overground gait training, and gait training with the study device. Rest periods will be provided as necessary during the training visits.

SUMMARY:
The investigator plans to test the use of the Ekso Bionics® Gait Training (Ekso GT™) exoskeleton for gait training in MS patients. The device will solely be used in the clinic under direct supervision from a physical therapist. This is a small PI-initiated uncontrolled pilot study to gather safety and feasibility data on the exoskeleton in individuals with MS and walking impairment.

DETAILED DESCRIPTION:
Powered exoskeletons are approved by the FDA to assist in the rehabilitation of persons with spinal cord injury and post-stroke hemiplegia. The investigator is aware of only one pilot study of a powered exoskeleton (ReWalk®) in multiple sclerosis (MS) which demonstrated some improvements in sitting, standing and walking posture when used consistently. The investigator is not aware of any study of the Ekso GT™ exoskeleton in MS.

This is a feasibility and safety study of using the Ekso GT™ exoskeleton for gait training in patients with relapsing or progressive MS and severe mobility limitations (EDSS 5-5 - 7.5). Preliminary efficacy outcomes on gait and walking will also be collected for the purpose of designing a larger clinical trial of the Ekso GT™ exoskeleton for gait training in patients with MS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MS per 2017 revised McDonald criteria
* EDSS score 5.5-7.5 (moderate to severe walking disability)
* Cleared for gait training with the study device by the study treating physician

Device-Specific Criteria

* Involved in a standing program or must be able to tolerate at least 15 min upright without signs or symptoms of orthostatic hypotension
* Weigh 220 pounds (100kg) or less
* Be able to fit into the Ekso device:
* Between approximately 5'0" and 6'4" tall (really depends on leg measurements)
* Sufficient diaphragmatic strength such that respiration is not compromised with exercise

Assessed by physical therapy:

* Standing hip width of approximately 18" or less
* Have near normal range of motion(ROM) in hips, knees and ankles
* Sufficient upper extremity strength to use a front wheeled walker by manual muscle testing (minimum triceps strength bilaterally of 3/5, shoulder abduction and flexion/extension of 4/5 OR as discussed during demo, 2 normally functioning limbs such as in hemiplegia)

Exclusion Criteria:

* • MS exacerbation, severe acute comorbidity or surgery less than 90 days prior to enrollment

  * Diagnosed with osteoporosis or history of long bone fractures since diagnosis
  * Safety concern due to neurologic impairments (e.g. upper extremity weakness, visual loss) or comorbidities (e.g. cardiac, respiratory)
  * Other neurologic or non-neurologic condition interfering with walking
  * < 1 month since previous intensive gait training regimen or initiation of treatment that can affect walking (e.g. medication for spasticity)
  * Planned change in medications that may affect walking during the study period
  * Uncontrolled or severe orthostatic hypotension that limits standing tolerance
  * Active heterotrophic ossification (HO), hip dysplasia, or uncontrolled hip/knee axis abnormalities
  * Score <22 on the Mini-Mental State Examination or deemed to have cognitive impairment precluding safe training with the device during the screening and training process
  * Colostomy
  * Pregnancy
  * Unresolved deep vein thrombosis
  * Uncontrolled autonomic dysreflexia
  * Currently involved in another rehabilitation study

Assessed by physical therapy:

* Severe spasticity that prevents joint motion (severe stiffness or rigidity) in proximal lower extremity muscles, including hip adductors and knee flexors/extensors.
* Hip flexion contracture greater than ~17°
* Knee flexion contracture greater than 12°
* Unable to achieve neutral ankle dorsiflexion with passive stretch (achieve neutral with up to 12° knee flexion)
* Leg length discrepancy greater than 0.5" for upper leg, greater than 0.75" for lower leg
* Spinal instability
* Severe muscular or skeletal pain
* Open skin ulcerations on buttocks or other body surfaces in contact with exoskeleton or harness
* Shoulder extension range of motion(ROM) < 50° excludes using crutches during sit to stand or vice versa. (Walking with crutches permitted, sit <> stand would be done with walker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-07-23 (Actual); Primary Completion 2020-01-09 (Actual); Study Completion 2020-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francois A Bethoux, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Neurological Institute Mellen Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited and enrolled between July 2019 and October 2019 in the outpatient clinic.
Period: Overall Study
Arm/Group | Gait Training With Exoskeleton Device
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Gait Training With Exoskeleton Device
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 3
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 5
The Expanded Disability Status Scale = 5.5 to 7.5.Range from 0 to 10, higher scores worse outcome [Mean (Standard Deviation); unit: units on a scale] — The Expanded Disability Status Scale (EDSS) is a comprehensive, quantitative neurological examination, and is the most widely used measure of MS-related disability for clinical and research purposes. Scores range from 0 to 10, with higher scores representing a worse outcome.
  units on a scale | 6.30 (0.27)

OUTCOME MEASURES:

1. Primary Outcome: Dropout Rate
Description: Percentage of enrolled participants who drop out of the study before the end of the treatment period.
Time Frame: 0-14 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Gait Training With Exoskeleton Device
Number analyzed (Participants) | 5
Participants | 0

2. Primary Outcome: Adverse Events
Description: .All adverse events were collected throughout the study for each participant, up to 14 weeks",
Time Frame: 0-14 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Gait Training With Exoskeleton Device
Number analyzed (Participants) | 5
Participants | 4

3. Secondary Outcome: Timed 25 Foot Walk
Description: Change in walking speed on the Timed 25 Foot Walk between baseline, end of treatment, and end of follow-up period.
Time Frame: 0-14 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Gait Training With Exoskeleton Device
Number analyzed (Participants) | 5
seconds
  Baseline to end of treatment | 0.72 (1.20)
  Baseline to end of follow-up | 1.24 (2.87)

ADVERSE EVENTS:
Time Frame: all adverse events were collected throughout the study for each participant, up to 14 weeks.
Description: All probable and possibly related to device use events were collected along with other adverse events including falls
Arm/Group | Gait Training With Exoskeleton Device
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 4/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gait Training With Exoskeleton Device (N=5)
Fall (Nervous system disorders) | 2 (2) — None of the falls occurred during treatment visits.
Low back pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Chest wall soreness (Musculoskeletal and connective tissue disorders) | 1 (1) — Subsequent to a fall
Skin abrasion (Skin and subcutaneous tissue disorders) | 1 (1)
Back muscle weakness (Nervous system disorders) | 1 (1) — assessed as related to MS
Bruising (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-17): https://cdn.clinicaltrials.gov/large-docs/73/NCT04000373/Prot_SAP_001.pdf